CLINICAL TRIAL: NCT02253056
Title: Montag Ist Fasten-Tag (German) - MIFT [Monday is Fasting Day]
Brief Title: Monday is Fasting Day - Non-Randomized Trial on Intermittent Fasting
Acronym: MIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Immanuel Hospital, Berlin, Germany (Unknown)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIFT-Trial
Record Dates: First submitted 2014-09-19; First posted 2014-10-01 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Fasting; Caloric Restriction; Focus is to observe effects of fasting in healthy volunteers.
MeSH Terms: conditions — Fasting | interventions — Caloric Restriction; Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fasting (Experimental): Intermittent fasting over 8 weeks (one day per week)
  Interventions: Other: Fasting / Caloric Restriction
- Healthy diet (Active Comparator): Regular healthy diet according to current German (DGE) guidelines for healthy nutrition.
  Interventions: Other: Healthy Diet

INTERVENTIONS:
Other: Fasting / Caloric Restriction
  Arms: Fasting
Other: Healthy Diet
  Arms: Healthy diet

SUMMARY:
The aim of this pilot study is to evaluate the effects of one regular fasting day per week over a total period of 8 weeks compared to a normal-eating habits among healthy volunteers.

DETAILED DESCRIPTION:
Participants in the intervention group receive an initial group training for fasting. Then all participants will observe one fixed fasting day per week (monday) over a total period of eight weeks.

Participants in the control group receive an initial group training for healthy diet according to current German guidelines (DGE). Moreover, they will receive the same offer as in the intervention group at the end of the 8-week study period. Until then the control group participants follow a regular healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* age 18 -65 yrs
* written informed consent

Exclusion Criteria:

* severe chronic comorbidity
* eating disorders
* pregnancy
* planed pregnancy
* simultaneous participation in other trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Insulin-like growth factor 1 and brain-derived neurotrophic factor | Baseline and after 8 weeks
  Measurement of changes after 8 weeks

SECONDARY OUTCOMES:
Quality of life questionnaire: WHO-5 | Baseline, 8 weeks, 6 month
  Questionnaire
Profile of mood states questionnaire: POMS | Baseline, 8 weeks, 6 month
  Questionnaire
Anxiety and depression questionnaire: HADS | Baseline, 8 weeks, 6 month
  Questionnaire
Flourishing questionnaire | Baseline, 8 weeks, 6 month
  Questionnaire
Visual analogue scales and Likert-scales | Baseline, 8 weeks, 6 month
  Questionnaire
Body Impedance Analysis (BIA) | Baseline, 8 weeks
  Measurement of changes after 8 weeks
Body weight and abdominal circumference | Baseline, 8 weeks
  Measurement of changes after 8 weeks
Systolic and diastolic bloodpressure | Baseline, 8 weeks
  Measurement of changes after 8 weeks
Blood: total cholesterol, LDL, HDL, Triglycerides; Insulin, GOT,GPT, GGT, AP; HbA1c; PTT, INR | Baseline and 8 weeks
  Changes after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, MD, Principal Investigator — Charité Medical University
Locations (1):
- Immanuel Hospital Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Research Institute´s Homepage — http://www.naturheilkunde.immanuel.de